CLINICAL TRIAL: NCT03753360
Title: Immunological and Genomic Effects of an Online Mindfulness Program for Stress Management
Brief Title: Online Mindfulness Program for Stress Management
Acronym: IGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Leonard Calabrese, Director of the RJ Fasenmyer Center for Clinical Immunology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-681
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Stress, Psychological; Burnout, Professional
Keywords: Stress; Mindfulness; Meditation; Gene expression; Immune; Online; Healthcare workers; Burnout; Cytokines; Cortisol
MeSH Terms: conditions — Stress, Psychological; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Prospective Parallel non-blinded randomized two arms, intervention group and active control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): internet-based mindfulness meditation program
  Interventions: Behavioral: Internet-Based Mindfulness Program - Stress Free Now for Healers
- Active Control Group (Other): relaxing music
  Interventions: Behavioral: Active Control Group - Relaxing Music

INTERVENTIONS:
Behavioral: Internet-Based Mindfulness Program - Stress Free Now for Healers — Stress Free Now for Healers is an online stress management program developed at Cleveland. It's delivered in 4 components:1Weekly introductions to the concepts and meditation theme are delivered via Web page views or a 5to10-min audio clip2Weekly guided meditations 5-20 min ea.available as embedded/downloadable mp3 on the website or via the Stress Free Now for Healers phone app,which participants are invited to practice at least 4 times each week and to record those practices3Daily articles provide the scientific underpinnings and merits of each week's theme or discuss various cognitive and behavioral strategies,activities,and concepts supporting or related to mindfulness4Daily tips suggesting how to manage stress or incorporate mindfulness in daily activities,including motivational quotes.Participants will have access to a smartphone app with recordings of the 11 guided meditations.Ea. participant will be assigned an e-coach that will communicate with the participant at least weekly.
  Arms: Intervention Group
Behavioral: Active Control Group - Relaxing Music — The control group will be given a flash drive and a link to a website where they can download several digital recordings of relaxing music and will be instructed to quietly listen to one or more of the recordings for at least 5 minutes every day for 6 weeks.
  Arms: Active Control Group

SUMMARY:
This is a prospective parallel non-blinded randomized study with two arms, an intervention group and an active control group.

Sixty healthy, but stressed nurses will be randomly assigned to either participate in a 6-week internet-based mindfulness meditation program produced by the Cleveland Clinic called Stress Free Now for Healers or to listen to relaxing music for at least 5 minutes a day for 6 weeks, and pre-post comparisons will be made for RNA expression profiles, plasma cytokine concentrations, telomerase activity, 6-point salivary cortisol and several self-reported assessments of physical and mental health.

DETAILED DESCRIPTION:
Chronic psychological stress is becoming increasingly pervasive in modern society, with 59% of working age adults who seek primary health care for any reason suffering from significant levels of stress. With long work hours and every increasing demands, healthcare workers are at an especially high risk of experiencing excessive amounts of stress, with over 50% of U.S. physicians and 34% of nurses now reporting symptoms of burnout. Psychological stress has been shown to have a variety of detrimental effects on the immune system, including an increased susceptibility to infection, a diminished immune response to vaccines, reactivation of chronic infections, and the development of chronic inflammation, which in turn is a contributing factor to the development and exacerbation of a wide variety of chronic conditions. Acute stress activates the hypothalamic-pituitary-adrenal (HPA) axis and the sympathetic nervous system, provoking the release of various hormones such as ACTH, cortisol, and catecholamines, which in turn alter the functions of immune cells and generally lead to increased production of inflammatory cytokines, including, IL-6, IL-1β, IL-10, and TNF-α . The communication between the neuroendocrine system and the immune system is bidirectional as cytokines also influence hormone production and the brain's response to stress. When experienced acutely, this physiologic response is harmless. However, when the stress is chronic it can lead to dysregulation of the immune system, setting the individual up for a host of problems ranging from serious infections to chronic inflammatory diseases like rheumatoid arthritis, heart disease, Alzheimer's and overall accelerated aging.

Various strategies have been used to counteract both the psychological and physiological effects of chronic stress including cognitive behavioral therapy, yoga, meditation, biofeedback, and others. While all of these have shown benefits, meditation, in particular, has recently gained widespread popularity as a simple and effective intervention for reducing stress. An ancient practice associated with many religions and cultures in different forms, meditation generally involves a calm and relaxed state of focus or concentration. Although its purpose has historically been to help the practitioner gain spiritual insight and achieve some form of enlightenment, it is now being studied as a way to improve mental and physical health. The most extensively studied form of meditation in the medical literature is the 8-week Mindfulness-Based Stress Reduction (MBSR) program developed by Jon Kabat Zinn, which has been shown to benefit patients with a wide variety of mental and physical health conditions.

One mechanism by which this and other forms of meditation are thought to exert their beneficial effects is through their anti-inflammatory effects, affecting the immune system at the cellular and molecular level. For example, a randomized controlled trial in older adults that went through the 8-week MBSR course showed a more than 25% pre-post change in 143 genes, including reduced activity of NF-kB target genes, relative to controls. But, similar changes have been observed in less time-intensive programs. Just 12 minutes a day of Kirtan Kriya Meditation for 8 weeks led to changes in 63 genes in a group of dementia caregivers compared to those who only listened to relaxing music. The observed changes included downregulation of inflammatory cytokines and NF-kB related transcripts as well as upregulation of immunoglobulin-related transcripts and interferon response factors.Some changes may even occur in as little as one day. Kaliman and colleagues showed that following an 8-hour meditation retreat experienced meditators showed reduced expression of histone deacetylases, global histone modifications, and downregulation of pro-inflammatory genes compared to a group of non-meditators who spent the same time simply relaxing. A meta-analysis of randomized trials has also shown consistently positive effects of meditation on immune cell telomeres, which is a marker of immune cell aging. As Epel and colleagues recently showed, many of these effects may be due to a non-specific relaxation response, especially in novices.However, when Creswell and colleagues compared the changes in a group of stressed, unemployed adults that went through either a 3-day meditation retreat or a 3-day relaxation retreat at the same center, only the meditation group showed a sustained reduction in IL-6 that could be accounted for, in part, by connectivity changes within the brain.Two recent papers have done an excellent job of summarizing the current knowledge regarding the molecular signature associated with mind-body training, and the reader is referred to these for a more detailed review of the topic.

Despite their effectiveness, a major limitation of MBSR and similar programs is a formidable time commitment and a high dropout rate, limiting its utility as a practical intervention for stress management in the population at large, especially busy healthcare workers. It would be ideal to have a more scalable intervention which economizes on time, adapts to modern lifestyles and is inexpensive. Accordingly, the Cleveland Clinic developed an online mindfulness-based stress reduction program known as Stress Free Now. A 6-week program with short daily online articles with tips and ideas for reducing stress and an accompanying app with guided meditations, Stress Free Now is designed for the modern man or woman and capable of reaching the masses. In 2013, a study showed that participants in this program experienced significant stress reductions and improvement in other psychological measures compared to controls. What remains to be answered is whether this program will exhibit biological effects comparable to those seen with in-person interventions. This is the purpose of this project. Using whole transcriptome sequencing and measurement of circulating cytokines, telomerase activity, and diurnal cortisol rhythms the investigators plan to characterize the molecular and immunological phenotype associated with participating in an internet-based mindfulness meditation program. It is hypothesized that following participation in Stress Free Now for Healers, participants will exhibit downregulation of pro-inflammatory gene pathways as well as reduced circulating levels of inflammatory cytokines, increased telomerase activity and reduced, smoother diurnal cortisol patterns compared to controls. This knowledge would be significant because it would provide, for the first time, mechanistic evidence of the benefits of a brief, internet-based mindfulness-meditation program, supporting the implementation this and similar programs into clinical practice. The present study will be a prospective parallel non-blinded randomized study with two arms, an intervention group and an active control group.

In brief, 60 healthy healthcare workers will be randomly assigned to either participate in a 6-week internet-based mindfulness meditation program produced by the Cleveland Clinic called Stress Free Now for Healers or to listen to relaxing music for at least 5 minutes a day for 6 weeks, and pre-post comparisons will be made for RNA expression profiles, plasma cytokine concentrations, telomerase activity, 6-point salivary cortisol and several self-reported assessments of physical and mental health.

Procedure

A total of 60 healthy, but stressed nurses will be enrolled in this study. After being screened and providing consent to participate, all subjects will schedule an initial study visit with the study coordinator at Cleveland Clinic Main Campus between the hours of 6 am and 11 am. They will be asked to arrive to this visit having fasted for 8-12 hours prior.

Study Visit 1: Upon arrival, the consent form will be reviewed and signed by both the participant and the study coordinator, and a copy of the form will be provided to the participant for his or her records. Any questions the participant has regarding the study will also be answered at this time. The participant will then be asked a few questions regarding his or her medical history and current medications. The participant will then be asked to fill out several assessments regarding his or her mental, emotional and physical health. The participant will then have 3, 10 mL tubes and 1, 2.5 mL tube of blood drawn, after which the participant will be monitored for at least 5 minutes for signs of dizziness or lightheadedness. During this time, the study coordinator will inform the participant of his assignment and give instructions accordingly. If the participant has been assigned to the intervention group, the study coordinator will help register him or her for the Stress Free Now course and show him or her both how and where to access the website and download the app on his or her phone. The participant will be instructed to begin the program the day of his or her first study visit. If the participant has been assigned to the control group, the study coordinator will show him or her how to access the relaxing music recordings and instruct him or her to listen to one of the recordings for at least 5 minutes every day for the next 6 weeks. The participants in the control group will have access to the Stress Free Now course at no charge at the conclusion of the study.

Study Visit 2: The final study visit will be scheduled for a time between 6 am and 11 am within one week of the conclusion of the 6-week period from initial study visit. The participant will be again asked to fast for 8-12 hours prior to the study visit. Upon arrival, the participant's medical history and medications will be reviewed for any changes, and any questions the participant has will be answered. The participant will then be asked to fill out the same assessments that were administered during the initial study visit. Again, 3, 10 mL tubes and 1, 2.5 mL tube of blood will be drawn and the participant will be monitored for at least 5 minutes for signs of dizziness or lightheadedness. The participant will then be thanked for participating in the study and provided with the agreed upon compensation. The participant will also be told to look out for an email in 6 weeks with a link to the same questionnaires the participant filled out in the first and last study visits. If the participant does not complete the online questionnaires within 2 days of being emailed the link, the participant will be sent an email reminder. Additional email reminders will be sent 1 and 2 weeks after the original link was sent if the questionnaires have still not been completed by these dates.

Salivary cortisol/DHEA test: At both study visit 1 and 2 participants will be provided with the Adrenocortex Stress Profile with Cortisol Awakening Response kit from Genova Diagnostics free of charge and told to collect all samples the next day following the printed instructions included in the kit. They will then ship the samples along with a requisition form containing only their study ID number, the date and time to Genova Diagnostics according to the instructions in the kit using the included prepaid shipping label. Once the samples have been processed and analyzed, the results will be uploaded to a password-protected online research account at gdx.net, to which only the principle and co-investigators will have access. A MTA/Data Use agreement between the Cleveland Clinic and Genova Diagnostics is in process and will be fully executed before the start of the study and the participants will be informed that the data of this test will be shared with an outside company.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female CCF nurses
* Abbreviated perceived stress scale (PSS-4) ≥ 7
* English speaking
* No history of major chronic medical conditions and/or diseases
* Able to provide informed consent and comply with study protocol

Exclusion Criteria:

* Significant chronic medical condition and/or disease
* Smoking
* Pregnancy
* Current use of antidepressants or any other psychiatric medication
* Current diagnosis of anxiety and/or depression
* History of any psychiatric diagnosis other than anxiety or depression
* Estrogen or hormone replacement therapy use
* Diagnosis of post-traumatic stress disorder
* Current use of any immunosuppressive medication
* No current or past meditation practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Pre-/post-intervention changes in mRNA transcript abundance across the entire transcriptome of circulating immune cells in the intervention group relative to the control group. | 6 weeks
  Next Generation Sequencing (NGS) will be used to measure whole transcriptome RNA expression in peripheral blood mononuclear cells (PBMCs) of subjects before and after participation in Stress Free Now or the control intervention. This data will then be used to create a pre-post differential expression signature to identify genes that were significantly up- or downregulated across the entire group. The within group changes will then be compared between the intervention and the control group and analyzed for significant differences.
Pre-/post-intervention changes in IL-6 | 6 weeks
  Measure plasma concentrations of IL-6 before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.
Pre-/post-intervention changes in IL-8 | 6 weeks
  Measure plasma concentrations of IL-8 before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.
Pre-/post-intervention changes in IL-10 | 6 weeks
  Measure plasma concentrations of IL-10 before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.
Pre-/post-intervention changes in TNF-α | 6 weeks
  Measure plasma concentrations of TNF-α before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.
Pre-/post-intervention changes in IFN-γ | 6 weeks
  Measure plasma concentrations of IFN-γ before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.
Pre-/post-intervention changes in peripheral blood mononuclear cell (PBMC) telomerase activity | 6 weeks
  Measure telomerase activity in PBMCs before and after participation in Stress Free Now for Healers or the control intervention and compare the change over time between groups.

SECONDARY OUTCOMES:
Pre-/post-intervention changes in salivary cortisol awakening response | 6 weeks
  The pre/post-changes in cortisol awakening response, measured via subject-collected saliva samples immediately upon and 30 minutes after waking, will be compared between groups.
Pre-/post-intervention changes in evening salivary cortisol | 6 weeks
  The pre/post-changes in evening cortisol level, measured via subject-collected saliva samples between 10 PM and 12 AM, will be compared between groups.
Pre-/post-intervention changes in diurnal cortisol slope | 6 weeks
  The pre/post-changes in diurnal cortisol slope, measured via subject-collected saliva samples at 6 time points throughout the day, will be compared between groups.
Pre-/post-intervention changes in perceived stress | 6 and 12 weeks
  The pre/post-changes in perceived stress, measured with a validated survey (Perceived Stress Scale), will be compared between groups. The Perceived Stress Scale is a 10-item scale with a total score ranging between 0 and 40 used to measure of the degree to which situations in one's life are appraised as stressful. A higher score indicates a higher level of perceived stress.
Pre-/post-intervention changes in resilience | 6 and 12 weeks
  The pre/post-changes in psychological resilience, measured with a validated survey (Connor-Davidson Resilience Scale abbreviated version), will be compared between groups. The Connor-Davidson Resilience Scale abbreviated version is 10-item scale that measures psychological resilience using a total score between 0 and 40, with a higher score indicating greater resilience.
Pre-/post-intervention changes in symptoms of burnout | 6 and 12 weeks
  The pre/post-changes in symptoms of professional burnout, measured with a validated survey (Maslach Burnout Inventory - Human Services Survey), will be compared between groups. The Maslach Burnout Inventory - Human Services Survey is the original and most widely used version of the Maslach Burnout Inventory and is designed to measure symptoms of work-related burnout in professionals of human services. It is a 22-item scale that gives a total score ranging between 0 and 132, with higher scores indicating the respondent experiencing more burnout.
Pre-/post-intervention changes in emotional well-being | 6 and 12 weeks
  The pre/post-changes in emotional well-being, measured with a validated survey (RAND 36 - Emotional Well-Being subscale), will be compared between groups.
Pre-/post-intervention changes in self-reported global health | 6 and 12 weeks
  The pre/post-changes in global health, measured with a validated survey (PROMIS Global Health SF), will be compared between groups. The PROMIS Global Health Short Form is a 10-item scale used to assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life, with the total score ranging between 10 and 50, higher scores indicating greater overall health.
Pre-/post-intervention changes in anxiety symptoms | 6 and 12 weeks
  The pre/post-changes in anxiety, measured with a validated survey (PROMIS Anxiety CAT), will be compared between groups. The PROMIS Anxiety CAT is a computer adaptive test that measures anxiety related symptoms. For CATs, the number of items varies between 4 and 12. The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. The CAT will continue until either the standard error drops below a specified level or the participant has answered the maximum number of questions (12), whichever occurs first. The end result is a T-score in which the individual's responses are compared to the U.S. general population, which based on calibration testing has a mean of 50 and a standard deviation of 10. A higher score indicates higher levels of anxiety.
Pre-/post-intervention changes in depressive symptoms | 6 and 12 weeks
  The pre/post-changes in depressive symptoms, measured with a validated survey (PROMIS Depression CAT), will be compared between groups. The PROMIS Depression CAT is a computer adaptive test that measures anxiety related symptoms. For CATs, the number of items varies between 4 and 12. The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. The CAT will continue until either the standard error drops below a specified level or the participant has answered the maximum number of questions (12), whichever occurs first. The end result is a T-score in which the individual's responses are compared to the U.S. general population, which based on calibration testing has a mean of 50 and a standard deviation of 10. A higher score indicates higher levels of depression.
Pre-/post-intervention changes in fatigue | 6 and 12 weeks
  The pre/post-changes in fatigue, measured with a validated survey (PROMIS Fatigue CAT), will be compared between groups. The PROMIS Fatigue CAT is a computer adaptive test that measures anxiety related symptoms. For CATs, the number of items varies between 4 and 12. The response to the first item will guide the system's choice of the next item for the participant. The participant's response to the second item will dictate the selection of the following question, and so on. The CAT will continue until either the standard error drops below a specified level or the participant has answered the maximum number of questions (12), whichever occurs first. The end result is a T-score in which the individual's responses are compared to the U.S. general population, which based on calibration testing has a mean of 50 and a standard deviation of 10. A higher score indicates higher levels of fatigue.
Pre-/post-intervention changes in sleep quality | 6 weeks
  The pre/post-changes in sleep quality, measured with a validated survey (Insomnia Severity Index), will be compared between groups. The Insomnia Severity Index is a 7-item scale with a total score ranging between 0 and 28 that is used to assess the level of subjective sleep difficulties and insomnia-related symptoms over the past 2 weeks. A higher score indicates reduced sleep quality and more insomnia-related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860